CLINICAL TRIAL: NCT02488785
Title: The Impact of a Comprehensive Virtual Diabetes Self-Care and Education Program on Diabetes-related Outcomes in Latinos With Type 2 Diabetes
Brief Title: Impact of a Virtual Diabetes Self-Care and Education Program on Diabetes-related Outcomes in Latinos With T2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Joslin Diabetes Center (Other)
Collaborators: Verizon Foundation (Other); DHR Health Institute for Research and Development (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014-42
Record Dates: First submitted 2015-06-04; First posted 2015-07-02 (Estimated); Results first posted 2022-09-06 (Actual); Last update posted 2022-09-06 (Actual); Status verified 2022-08

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Type 2 Diabetes Mellitus; Telehealth; Hispanics; Latinos; Self-Care; Mobile Health; mHealth
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): Patients in this group will attend regular clinical and education appointments as offered by the clinic for their diabetes care.
- Intervention (Experimental): Patients in this group will be part of a Virtual Diabetes Self-Care and Education Program. They will receive a phone to communicate with a diabetes educator for 6 months. They will connect with the diabetes educator for weekly video conferences of up to 30 minutes for twelve consecutive weeks, followed by 7 phone calls. Additionally, they will receive a weekly text message about diabetes for 6 months.
  Interventions: Behavioral: Virtual Diabetes Self-Care and Education Program; Device: Fitbit; Device: Smartphone

INTERVENTIONS:
Behavioral: Virtual Diabetes Self-Care and Education Program — Participants will be able to have frequent contact in order to share physical activity and glucose data with the diabetes educator using the smartphone they will receive. Information downloaded to the Glooko Population Management tool can be shared with the diabetes educator.
  Arms: Intervention
Device: Fitbit — Participants will be given a Fitbit physical activity tracker which they can use to record their activity and share the information with the diabetes educator using the device's smartphone application.
  Other Names: physical activity tracker
  Arms: Intervention
Device: Smartphone — All virtual visits were performed via provided smartphone. In addition, participants will receive a Glooko MeterSync Blue cable which is able to connect to most glucose meters in order to download glucose data to the Glooko Population Management tool on their smartphones
  Arms: Intervention

SUMMARY:
The goal of this study is to evaluate the impact of a comprehensive diabetes education and management program based on frequent communication with patients using teleconsultation, text messaging, and phone calls on diabetes related outcomes in Latino patients with type 2 diabetes. The investigators hypothesize that the decline in hemoglobin A1c value between the baseline and the six-month visit will be at least 0.5 percent greater in the intervention group than in the control group.

DETAILED DESCRIPTION:
In this study participants will be followed for a period of 9 months. The control group will receive usual care during this period of time. While, the intervention group will be part of a diabetes education and management program lasting 6 months via a smartphone participants will receive. The 6 month intervention will be followed by a 3 month observation period.

ELIGIBILITY:
Inclusion Criteria:

* Have physician-diagnosed type 2 diabetes
* Be self-identified as Hispanic or Latino
* An A1c value between 8-14% within the last three months.
* Demonstrate the ability, either alone or with the help of a family member that will be with the patient at least once a week, to use the technology that will be used during the teleconsultations

Exclusion Criteria:

* Severe diabetes related chronic complications such as chronic renal failure, blindness, amputations, stroke, etc.
* Concomitant chronic illnesses that would affect their participation in the program, i.e. cancer, debilitating diseases, etc.
* Any other condition that would affect participant's basic mental health skills
* Type 1 diabetes or gestational diabetes
* Patients with abnormal hemoglobin, anemia or any condition that may affect red blood cell turnover. Any of these conditions may be detected through participants' history or through the laboratory report at study screening
* Signs or symptoms of metabolic decompensation (polyuria, polydypsia, polyphagia, unexplained weight loss, blurry vision, lethargy, etc.)

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2017-03-31 (Actual); Study Completion 2017-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sylvia E Rosas, MD, Principal Investigator — Joslin Diabetes Center; Marcel Twahirwa, MD, Principal Investigator — Doctors Hospital at Reinassance
Locations (1):
- Doctors Hospital at Renaissance, Edinburg, Texas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention: Patients in this group will be part of a Virtual Diabetes Self-Care and Education (DSME) Program. They will receive a phone to communicate with a diabetes educator (DE) for 6 months. They will connect with the DE for weekly video conferences of up to 30 minutes for twelve consecutive weeks, followed by 7 phone calls. They will receive a weekly text message about diabetes for 6 months.
  Virtual (DSME) Program: Participants will have frequent contact in order to share physical activity and glucose data with the DE using the smartphone they will receive. Information downloaded to the Glooko Population Management tool can be shared with the DE.
  Fitbit: Participants will be given a Fitbit physical activity tracker which they can use to record their activity and share the information with the diabetes educator using the device's smartphone application.
  Smartphone: All virtual visits were performed via provided smartphone. Participants will receive a Glooko MeterSyn
Period: Overall Study
Arm/Group | Control | Intervention
Started | 47 | 49
Completed | 41 | 38
Not Completed | 6 | 11

BASELINE CHARACTERISTICS:
Groups:
- Intervention: Patients (pt) in this group will be part of a Virtual Diabetes Self-Care and Education (DSME) Program. Pt will receive a phone to connect with a diabetes educator (DE) for 6 months. Pt will have a weekly video call of up to 30 min. with the DE for 12 weeks, followed by 7 phone calls. Pt will get a weekly text message about diabetes for 6 months.
  Virtual DSME Program: pt will have frequent contact in order to share physical activity and glucose data with the DE using smartphone. Information downloaded to the Glooko can be shared with the DE.
  Fitbit: Participants will be given a Fitbit physical activity tracker which they can use to record their activity and share the information with the DE using the device's smartphone application.
  Smartphone: All virtual visits were performed via. In addition, pt will receive a Glooko MeterSync which is able to connect to most glucose meters in order to download glucose data to the Glooko Population Management tool on their smartphones
- Total: Total of all reporting groups
Arm/Group | Control | Intervention | Total
Number analyzed (Participants) | 47 | 49 | 96
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.6 (11.5) | 50.9 (11.8) | 54.2 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 29 | 61
  Male | 15 | 20 | 35
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 47 | 49 | 96
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 47 | 49 | 96
Hemoglobin A1C [Mean (Standard Deviation); unit: %] | 9.56 (1.3) | 9.97 (1.78) | 9.7 (1.5)

OUTCOME MEASURES:

1. Primary Outcome: Hemoglobin A1c
Description: The A1C test is a blood test used to diagnose type 2 diabetes and then to manage diabetes. It is measured as a percent.
Time Frame: 9 months
Measure: Mean (Standard Deviation); unit: percentage of A1C
Arm/Group | Control | Intervention
Number analyzed (Participants) | 39 | 36
percentage of A1C | 8.41 (1.55) | 8.18 (1.59)

ADVERSE EVENTS:
Time Frame: We did not collect any adverse events as this was a behavioral intervention that did not modify standards of care
Description: While we did not monitor for mortality, there were no reports of patient death during the study period.
  Serious adverse events were not monitored. Other adverse events were not monitored.
Groups:
- Intervention: Patients in this group will be part of a Virtual Diabetes Self-Care and Education (DSME) Program. They will receive a phone to communicate with a diabetes educator for 6 months. They will connect with the diabetes educator for weekly video conferences of up to 30 minutes for twelve consecutive weeks, followed by 7 phone calls. Additionally, they will receive a weekly text message about diabetes for 6 months.
  Virtual (DSME) Program: Participants will be able to have frequent contact in order to share physical activity and glucose data with the diabetes educator using the smartphone they will receive. Information downloaded to the Glooko Population Management tool can be shared with the diabetes educator.
  Fitbit: Participants will be given a Fitbit physical activity tracker which they can use to record their activity and share the information with the diabetes educator using the device's smartphone application.
  Smartphone: All virtual visits were performed vi
Arm/Group | Control | Intervention
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-10-27): https://cdn.clinicaltrials.gov/large-docs/85/NCT02488785/Prot_SAP_000.pdf